CLINICAL TRIAL: NCT00367211
Title: A 6-Month, Phase 3, Randomized, Double-Blind, Parallel-Group, Controlled, Multi-Center Study to Evaluate the Incidence of Gastric Ulcers Following Administration of Either PN 200 or Naproxen in Subjects Who Are at Risk for Developing NSAID-Associated Ulcers.
Brief Title: Study to Evaluate the Incidence of Gastric Ulcers Following Administration of Either PN 200 or Naproxen in Subjects Who Are at Risk for Developing NSAID-Associated Ulcers.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: David Taylor, Pozen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PN200-301
Expanded Access: Available
Record Dates: First submitted 2006-08-18; First posted 2006-08-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Ankylosing Spondylitis
Keywords: Gastric Ulcers; NSAID; Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Stomach Ulcer; Arthritis | interventions — Naproxen; Omeprazole

INTERVENTIONS:
Drug: PN 200 tablets (500 mg naproxen and 20 mg omeprazole)
Drug: Naproxen 500 mg tablets (PN 200 minus omeprazole)

SUMMARY:
The purpose of this study is to evaluate the incidence of gastric ulcers following administration of either PN 200 or Naproxen in subjects who are at risk for developing NSAID-associated ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female subjects with a history of osteoarthritis, rheumatoid arthritis, ankylosing spondylitis or other medical conditions expected to require daily NSAID therapy for at least 6 months who are 18-49 years of age and have a history of a documented, uncomplicated gastric or duodenal ulcer (a mucosal break of at least 3 mm in diameter with depth, without any concurrent bleeding, clot or perforation) within the past 5 years OR, who are 50 years of age and older (these subjects do not require a history of a documented, uncomplicated gastric or duodenal ulcer within the past 5 years).
* Female subjects are eligible for participation in the study if they are of:

  1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant); or,
  2. Childbearing potential, have a negative pregnancy test (urine) at screening, and at least one of the following applies or is agreed to by the subject:

     * Complete abstinence from intercourse for at least 14 days prior to first dose of study drug, throughout the study, and for 30 days after completion of the study
     * Female sterilization or sterilization of male partner; or,
     * Hormonal contraception by oral route, implant, injectable, vaginal ring; or,
     * Any intrauterine device (IUD) with published data showing that the lowest expected failure rate is less than 1% per year;
     * Double barrier method (2 physical barriers or 1 physical barrier plus spermicide); or
     * Any other method with published data showing that the lowest expected failure rate is less than 1% per year.
* Each subject must be able to understand and comply with study procedures required of a subject and is able and willing to provide written informed consent prior to any study procedures being performed.

Exclusion Criteria:

* History of hypersensitivity to omeprazole or to another proton-pump inhibitor.
* History of allergic reaction or intolerance to any NSAID (including aspirin) and/or subject has a history of NSAID-induced symptoms of asthma, rhinitis, and/or nasal polyps.
* Participation in any study of an investigational treatment in the 4 weeks before screening.
* Presence of uncontrolled acute or chronic medical illness, e.g. gastrointestinal disorder, diabetes, hypertension, thyroid disorder, depression and/or infection that would endanger a subject if they were to participate in the study.
* Gastrointestinal disorder or surgery leading to impaired drug absorption.
* Evidence of uncontrolled, or unstable cardio- or cerebrovascular disorder, which in the investigator's opinion would endanger a subject if they were to participate in the study.
* Schizophrenia or bipolar disorder.
* Use of any excluded concomitant medication (see Section 9.2).
* A recent history (in the past 3 months) suggestive of alcohol or drug abuse or dependence, including overuse/abuse of narcotics for management of pain.
* Serious blood coagulation disorder including use of systemic anticoagulants.
* Positive test result for H. pylori at screening.
* Baseline endoscopy showing any gastric or duodenal ulcer at least 3 mm in diameter with depth.
* Screening laboratory value for ALT, AST >2 times the upper limit of normal.
* Estimated creatinine clearance < 30 ml/min.
* Other than noted specifically, any screening laboratory value that is clinically significant in the investigator's opinion and would endanger a subject if they were to participate in the study.
* History of malignancy, treated or untreated, within the past 5 years, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is the incidence of gastric ulcers, defined as a mucosal break of at least 3 mm in diameter (measured by close application of open endoscopic biopsy forceps) with depth, at anytime throughout 6 months of study treatment.

SECONDARY OUTCOMES:
The secondary efficacy variable is the incidence of duodenal ulcers at any time throughout 6 months of treatment, tolerability and safety.

CONTACTS AND LOCATIONS:
Locations (1):
- Patient Interaction, Pompano Beach, Florida, United States